CLINICAL TRIAL: NCT04312243
Title: Nitric Oxide Gas Inhalation for Prevention of COVID-19 in Healthcare Providers
Brief Title: NO Prevention of COVID-19 for Healthcare Providers
Acronym: NOpreventCOVID
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID wave passed and we closed the study prematurely
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NOpreCOVID-19
Record Dates: First submitted 2020-03-15; First posted 2020-03-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Coronavirus Infections; Healthcare Associated Infection
MeSH Terms: conditions — Coronavirus Infections; Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Inhaled NO (160 ppm) before and after the work shift. Daily monitoring of body temperature and symptoms. SARS-CoV-2 RT-PCR test if fever or COVID-19 symptoms.
  Interventions: Drug: Inhaled nitric oxide gas
- Control Group (No Intervention): Daily monitoring of body temperature and symptoms. SARS-CoV-2 RT-PCR test if fever or COVID-19 symptoms.

INTERVENTIONS:
Drug: Inhaled nitric oxide gas — Control group: a SARS-CoV2 rt-PCR will be performed if symptoms arise. Treatment group: the subjects will breathe NO at the beginning of the shift and before leaving the hospital. Inspired NO will be delivered at 160 parts per million (ppm) for 15 minutes in each cycle. A SARS-CoV-2 rt-PCR will be performed if symptoms arise. Safety: Oxygenation and methemoglobin levels will be monitored via a non-invasive CO-oximeter. If methemoglobin levels rise above 5% at any point of the gas delivery, inhaled NO will be halvened. NO2 gas will be monitored and maintained below 5 ppm.
  Arms: Treatment Group

SUMMARY:
Thousands of healthcare workers have been infected with SARS-CoV-2 and contracted COVID-19 despite their best efforts to prevent contamination. No proven vaccine is available to protect healthcare workers against SARS-CoV-2.

This study will enroll 470 healthcare professionals dedicated to care for patients with proven SARS-CoV-2 infection. Subjects will be randomized either in the observational (control) group or in the inhaled nitric oxide group. All personnel will observe measures on strict precaution in accordance with WHO and the CDC regulations.

DETAILED DESCRIPTION:
In their efforts to provide care for patients with novel coronavirus (SARS-CoV-2) disease (COVID-19) infection, many healthcare workers around the globe exposed to SARS-CoV-2 got infected and died over the past two months. Quarantined nurses and physicians have become the norm in regions with COVID-19 patients, putting at risk the overall functionality of the regional healthcare system. Other than strict contact-precautions, no proven vaccination or targeted therapy is available to prevent COVID-19 in healthcare workers. Inhaled nitric oxide gas (NO) has shown in a small clinical study to have antiviral activity against a Coronavirus during the 2003 SARS outbreak. We have designed this study to assess whether intermittent inhaled NO in healthcare workers might prevent their infection with SARS-CoV-2.

Background: After almost two months of fight against COVID-19 infection, on February 24, more than 3,000 physicians and nurses were reported as contracting COVID-19 disease in Wuhan (China). Fatalities among those healthcare workers were reported to be related to SARS-CoV-2 infection. Implementation of strict contact protections for all healthcare personnel is essential to decrease and contain the risks of exposure. However, despite best efforts, dozens of thousands of healthcare providers have been quarantined for at least 14 consecutive days in Wuhan alone. Similarly data have been reported in Italy, several healthcare providers have been quarantined, developed pneumonia and died. Most recent information from Italy reported that 12% of healthcare workers are infected.

The shortage of hospital personnel, especially in the critical care and anesthesiology domains, led many hospitals to postpone indefinitely scheduled surgical procedures, including cardiac surgery or oncological procedures. Only urgent and emergent cases are performed in patients without symptoms (i.e., absence of fever, cough or dyspnea), no signs (i.e., negative chest CT for consolidations, normal complete blood count) and a negative test on SARS-CoV-2 reverse transcriptase (rt)-PCR. If time does not allow for thorough screening (i.e., after traumatic injury), such patients are considered to be infected and medical staff in the OR are fully protected with third degree protections (i.e., N95 masks, goggles, protective garments and a gown and double gloving).

Rationale. In 2004 in a collaborative study between the virology laboratory at the University of Leuven (Belgium), the Clinical Physiology Laboratory of Uppsala University (Sweden) and the General Airforce Hospital of China (Beijing, China), nitric oxide (NO) donors (e.g. S-nitroso-N-acetylpenicillamine) greatly increased the survival rate of infected eukaryotic cells with the coronavirus responsible for SARS (SARS-CoV-1), suggesting direct antiviral effects of NO. These authors suggest that oxidation is the antiviral mechanism of nitric oxide. A later work by Akerstrom and colleagues showed that NO or its derivatives reduce palmitoylation SARS-CoV spike (S) protein affecting its fusion with angiotensin converting enzyme 2. Furthermore, NO or its derivatives reduce viral RNA synthesis in the infected cells. Future in-vitro studies should confirm that NO donors are equally effective against SARS-CoV-2, as the current virus shares 88% of its genome with the SARS-CoV [3]. However, at present it is reasonable to assess that a high dose of inhaled NO might be anti-viral against SARS-CoV-2 in the lung. The virus is transmitted by human-to-human contact and occurs primarily via respiratory droplets from coughs and sneezes within a range of about 1.5 meters. The incubation period ranges from 1 to 14 days with an estimated median incubation period of 5 to 6 days according to the World Health Organization [1]. COVID-19 disease is mainly a respiratory system disease, but in the most severe forms can progress to impair also other organ function (i.e., kidneys, liver, heart). Nitric oxide gas inhalation has been successfully and safely used for decades (since 1990) in thousands of newborns and adults to decrease pulmonary artery pressure and improve systemic oxygenation.

Recently at the Massachusetts General Hospital, a high dose of inhaled NO (160 ppm) for 30 - 60 minutes was delivered twice a day to an adolescent with cystic fibrosis and pulmonary infection due to multi-resistant Burkholderia cepacia. There were no adverse events to this patient, blood methemoglobin remained below 5% and lung function and overall well-being improved.

Clinical Gap. Thousands of healthcare workers have been infected with SARS-CoV-2 and contracted COVID-19 despite their best efforts to prevent contamination. No proven vaccine is available to protect healthcare workers against SARS-CoV-2.

Hypothesis. Due to genetic similarities with the Coronavirus responsible for SARS, it is expected that inhaled NO gas retains potent antiviral activity against the SARS-CoV-2 responsible for COVID-19.

Aim. To assess whether intermittent delivery of inhaled NO gas in air at a high dose may protect healthcare workers from SARS-CoV-2 infection.

Observational group: daily symptoms and body temperature monitoring. SARS-CoV-2 RT-PCR test will be performed if fever or COVID-19 symptoms.

Treatment group: the subjects will breathe NO at 160 parts per million (ppm) for two cycles of 15 minutes each at the beginning of each shift and before leaving the hospital. Daily symptoms and body temperature monitoring. SARS-CoV-2 RT-PCR test will be performed if fever or COVID-19 symptoms. Safety: Oxygenation and methemoglobin levels will be monitored via a non-invasive CO-oximeter. If methemoglobin levels rise above 5% at any point of the gas delivery, inhaled NO will be stopped. NO2 gas will be monitored and maintained below 5 ppm.

Blinding. The treatment is not masked.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Scheduled to work with SARS-CoV-2 infected patients for at least 3 days in a week.

Exclusion Criteria:

1. Previous documented SARS-CoV-2 infections and subsequent negative SARS-CoV-2 rt-PCR test.
2. Pregnancy
3. Known hemoglobinopathies.
4. Known anemia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
COVID-19 diagnosis | 14 days
  Percentage of subjects with COVID-19 diagnosis in the two groups

SECONDARY OUTCOMES:
Positive SARS-CoV-2 rt-PCR test | 14 days
  Percentage of subjects with a positive test in the two groups

OTHER OUTCOMES:
Total number of quarantine days | 14 days
  Mean/ Median in the two groups
Proportion of healthcare providers requiring quarantine | 14 days
  Percentage in the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akerstrom S, Gunalan V, Keng CT, Tan YJ, Mirazimi A. Dual effect of nitric oxide on SARS-CoV replication: viral RNA production and palmitoylation of the S protein are affected. Virology. 2009 Dec 5;395(1):1-9. doi: 10.1016/j.virol.2009.09.007. Epub 2009 Oct 1. PMID 19800091
- [Background] Keyaerts E, Vijgen L, Chen L, Maes P, Hedenstierna G, Van Ranst M. Inhibition of SARS-coronavirus infection in vitro by S-nitroso-N-acetylpenicillamine, a nitric oxide donor compound. Int J Infect Dis. 2004 Jul;8(4):223-6. doi: 10.1016/j.ijid.2004.04.012. PMID 15234326
- [Derived] Akhtar S, Das JK, Ismail T, Wahid M, Saeed W, Bhutta ZA. Nutritional perspectives for the prevention and mitigation of COVID-19. Nutr Rev. 2021 Feb 11;79(3):289-300. doi: 10.1093/nutrit/nuaa063. PMID 33570583